CLINICAL TRIAL: NCT02977884
Title: Complete Health Improvement Program (CHIP) Risk Reduction/Claims Evaluation Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Touro University (Other)
Responsible Party: Principal Investigator, David Drozek, Assistant Professor, Ohio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12X81
Record Dates: First submitted 2016-11-18; First posted 2016-11-30 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Dyslipidemias; Overweight and Obesity
Keywords: nutrition; exercise; stress; cardiovascular disease; diabetes; hypertension; dyslipidemia; cholesterol; overweight; obesity; lifestyle
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Dyslipidemias; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Complete Health Improvement Program (Experimental): Participants in The Complete Health Improvement Program
  Interventions: Behavioral: The Complete Health Improvement Program

INTERVENTIONS:
Behavioral: The Complete Health Improvement Program — CHIP focuses on food, diet, activity, exercise, stress management, by viewing videos, cooking demonstrations, discussion, and exercise. Intervention nurtures intelligent self-care through enhanced understanding of the epidemiology, etiology, and risk factors associated with chronic lifestyle related diseases. The primary focus is the consumption of plant-based whole foods, such as fresh fruits, vegetables, whole grains, legumes, and nuts. The goal was to keep dietary fat below 20% of total calories, daily intake of added sugar below 10 tsps, sodium below 2,000 mg, and cholesterol below 50 mg. High fiber food intake (>35 g/day) is encouraged, and flexibility exercises, a daily walk of 30 minutes or 10,000 steps and daily use of stress management techniques.
  Other Names: CHIP

SUMMARY:
The project proposes to provide the Complete Health Improvement Program (CHIP) initially up to 25 adult (non-pregnant) Ohio University employees (and/ or their adult family members) with with diabetes / prediabetes, obesity / overweight, hypertension / prehypertension, atherosclerotic cardiovascular disease, or dyslipidemia in an effort to improve self-management and the consequences of biometric factors that can be modified by lifestyle changes. The CHIP program is an educationally based, lifestyle intervention program that aims to reduce healthcare cost, absenteeism, and increase employee productivity. The investigators expect that participants following the programs guidelines will lower their body mass index, cholesterol, reduce blood pressure and blood glucose levels, and therefore help to prevent chronic disease.

DETAILED DESCRIPTION:
In our Western culture, lifestyle changes focusing on diet, exercise and tobacco could prevent about 40% of all cancer deaths, and 82% of cardiac deaths, in the U.S. It is estimated that 71% of colon cancers, 70% of strokes, and 91% of diabetic cases could be avoided by living a healthy lifestyle. These health problems add a tremendous burden to our healthcare budget, and to the loss of productivity of our society. In 2007, it was estimated that 2.3 trillion dollars was spent on healthcare in the U.S., $7,600 for each individual. Expectations are that without dramatic change, this cost will continue to increase to unsustainable levels.

The Complete Health Improvement Program (CHIP) is a community based lifestyle medicine program with proven effectiveness in addressing these problems.

The project proposes to provide the Complete Health Improvement Program (CHIP) to adult (non-pregnant) Ohio University employees (and/ or their adult family members) with with diabetes / prediabetes, obesity / overweight, hypertension / prehypertension, atherosclerotic cardiovascular disease, or dyslipidemia in an effort to improve self-management and the consequences of biometric factors that can be modified by lifestyle changes. The CHIP program is an educationally based, lifestyle intervention program that aims to reduce healthcare cost, absenteeism, and increase employee productivity. The investigators expect that participants following the programs guidelines will lower their body mass index, cholesterol, reduce blood pressure and blood glucose levels, and therefore help to prevent chronic disease.

Ohio University Human Resources (HR) will provide research participants with scholarships to attend the CHIP program.

One aim of the project is to compare biometrics factors (weight, cholesterol, LDL, HDL, triglycerides, blood pressure, and fasting blood glucose, HgA1c) of participants before and after completion of the program (program completion defined as those who attended at least 14 of 16 CHIP classes, or 15 of the 18 new CHIP+ classes).

A second aim is to compare this groups health claims (health care utilization office visits, emergency room visits, hospitalizations, medication costs) with a control groups data (OU employees who have diabetes / prediabetes, obesity / overweight, hypertension / prehypertension, atherosclerotic cardiovascular disease, or dyslipidemia and do not participate in CHIP program).

A third aim is to compare the treatment groups absenteeism due to illness data with that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult, non-pregnant OU employees or adult families who are covered by Ohio University insurance and are participating in the Athens Complete Health Improvement Program

Exclusion Criteria:

* Pregnancy
* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Healthcare expenses | 2.5 years
  Healthcare costs

SECONDARY OUTCOMES:
Weight | 3 months
Fasting Glucose | 3 months
Fasting Lipid Profile | 3 months
Absenteeism: Sick days on record at Ohio University Human Resources | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: David S Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rankin P, Morton DP, Diehl H, Gobble J, Morey P, Chang E. Effectiveness of a volunteer-delivered lifestyle modification program for reducing cardiovascular disease risk factors. Am J Cardiol. 2012 Jan 1;109(1):82-6. doi: 10.1016/j.amjcard.2011.07.069. Epub 2011 Sep 23. PMID 21944675
- [Background] Leibold C, Shubrook JH, Nakazawa M, Drozek D. Effectiveness of the Complete Health Improvement Program in Reducing Risk Factors for Cardiovascular Disease in an Appalachian Population. J Am Osteopath Assoc. 2016 Feb;116(2):84-91. doi: 10.7556/jaoa.2016.020. PMID 26830523
- [Background] Vogelgesang J, Drozek D, Nakazawa M, Shubrook JH. Payer source influence on effectiveness of lifestyle medicine programs. Am J Manag Care. 2015 Sep 1;21(9):e503-8. PMID 26618437
- [Background] Drozek D, Diehl H, Nakazawa M, Kostohryz T, Morton D, Shubrook JH. Short-term effectiveness of a lifestyle intervention program for reducing selected chronic disease risk factors in individuals living in rural appalachia: a pilot cohort study. Adv Prev Med. 2014;2014:798184. doi: 10.1155/2014/798184. Epub 2014 Jan 16. PMID 24527219